CLINICAL TRIAL: NCT04542564
Title: Safety, Feasibility and Acceptability of Using TElemedicine to Replace Face-to-face Physician Consultation in Patients With HyperTension in Hong Kong: a Pilot Randomized-controlled Trial
Brief Title: TElemedicine to Replace Face-to-face Physician Consultation in Patients With HyperTension : a Pilot Randomized-controlled Trial
Acronym: SATE-HT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SATE-HT
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telemedicine group (Experimental): The HT app (HealthCap) allows patients to record their home BP measurements (HBPM) and can automatically provide mean BP values from the previous 7 or 30 days. 1-2 week prior to a scheduled physician, HealthCap and a research assistant will remind patients to take dual BP readings both in the morning and evening for 1 week for doctors' management. The mean values of the 7-day home BP will be checked before the index consultation. If the home BP control was optimal (i.e. ≤135/85 mmHg), other important parameters will be checked automatically by a questionnaire in the app: (i) if they have good drug compliance and if they experienced any side effects,(ii) if they have symptoms suggestive of target organ damages such as chest pain or hemiplegia, and (iii) if they have any problem(s) that need to consult a physician. If no complaints are identified, the patient can collect medications directly from the clinic and the physician appointment will be deferred for 3 months
  Interventions: Device: telemedicine; Other: usual care
- usual care (Placebo Comparator): Patients in the usual care group will be asked to refrain from downloading or using any health care apps related to HT
  Interventions: Other: usual care

INTERVENTIONS:
Device: telemedicine — a mobile app and telemedicine platform to confirm good blood pressure control and may save doctor face-to-face consultation
  Arms: telemedicine group
Other: usual care — These patients have unrestricted access to healthcare resources such as general outpatient clinics and emergency departments

SUMMARY:
The investigators has developed a blood pressure telemonitoring system. It is hypothesized that, when optimal control of BP is confirmed on the telemonitoring system, the index physician's consultation can be safely deferred, and medications can still be prescribed without such face-to-face consultation. Despite potentially resource-saving for doctors and time-saving for patients, the feasibility and patients' acceptability of the use of the telemonitoring system to replace face-to-face physician consultation remains unclear.

For primary outcome, the investigators hypothesize that this telemonitoring system will be feasible and acceptable to patients and can replace physicians' face-to-face consultations. For secondary outcomes, the investigators hypothesize that patients receiving care through telemonitoring have non-inferior BP control when compared with patients receiving usual care. Furthermore, the patients receiving telemonitoring may also have enhanced self-efficacy and compliance to drugs and lifestyle interventions

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of essential hypertension (HT) and are currently taking antihypertensive agents
* have good control of clinic BP as confirmed on ambulatory blood pressure monitoring (ABPM) (daytime BP ≤135/85mmHg)
* can read basic Chinese (as the content of the app in Chinese)
* have a home BP monitor (HBPM)
* used any mobile app (not HT-related) in the previous 1 year

Exclusion Criteria:

* an inability to give informed consent
* unwillingness to conduct HBPM or repeated ABPM
* current use of any other HT app for BP monitoring
* relative contraindications to ABPM (diagnosed atrial fibrillation, occupational drivers or patients with bleeding tendencies)
* severe mental illness, including those diagnosed with schizophrenia, dementia or as being actively suicidal, because these patients may have diminished ability to use the HT app;
* a diagnosis of other chronic disease(s) that need regular physical assessments and doctors' consultations (e.g. diabetes and asthma that are being treated, but patients with hypertension and hyperlipidaemia will remain eligible)
* diagnosed active cancer,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
rate of recruitment | baseline
  number of patients recruited per month during the recruitment period
rate of retention | baseline, 6-month
  number of dropouts during the 6-month study period
acceptability | at 6-month
  interview of around 20 patients in the intervention group

SECONDARY OUTCOMES:
blood pressure levels on 24-hour ambulatory blood pressure | baseline, 6-month
  daytime, nighttime, and 24-hour systolic and diastolic blood pressure
healthcare utilization | 6-month
  number of visits to general outpatient clinic, specialist clinic(s) and hospitalization during study period
self-efficacy scale | baseline, 6-month
  5-item self-efficacy scale specific to hypertension; a mean score from the items of a 9 or above were classified as having good self-efficacy
medication and diet adherence | baseline, 6-month
  Treatment Adherence Questionnaire for Patients with Hypertension (TAQPH); Score was summed to give a total range, higher score represented better adherence
exercise level | baseline, 6-month
  Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ); higher scores represented higher exercise level
eHealth literacy | baseline, 6-month
  Chinese 8-item eHealth literacy scale; higher scores represented higher eHealth literacy
health literacy | baseline, 6-month
  3-item Brief Health Literacy; higher scores represented higher health literacy

CONTACTS AND LOCATIONS:
Locations (1):
- Lek Yuen Clinic and Fanling clinic, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
May be available when inquired by other researchers

REFERENCES:
- [Derived] Wang S, Leung M, Leung SY, Han J, Leung W, Hui E, Mihailidou AS, Kam-Fai Tsoi K, Chi-Sang Wong M, Wong SY, Lee EK. Safety, Feasibility, and Acceptability of Telemedicine for Hypertension in Primary Care: A Proof-of-concept and Pilot Randomized Controlled Trial (SATE-HT). J Med Syst. 2023 Mar 11;47(1):34. doi: 10.1007/s10916-023-01933-4. PMID 36905441